CLINICAL TRIAL: NCT03569137
Title: Identification of Intestinal Microbiota Biomarkers Predictive of Diarrhea in Patients Treated by Ibrutinib.
Brief Title: Post-Ibrutinib Colitis and Intestinal Microbiota
Acronym: COLMI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Collaborators: Vendee Departmental hospital center (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC17_0463
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Gastrointestinal Microbiome
Keywords: Gut Microbiome; hematologic malignancies B; biomarkers; targeted therapy; Gut microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Identify gut microbiome biomarkers associated with colitis in patients treated with targeted therapy in hematology

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years
* Outside the context of guardianship, -affiliated to the Social Security Regime and
* Having consented to participate in the COLMI study.
* Patient who benefit of treatment by targeted therapy to Ibrutinib

Exclusion Criteria:

* History of uncontrolled colitis before the start of treatment.
* Patient with inflammatory bowel disease.
* Patient not consenting to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized in the Hematology departments and receiving targeted therapy with Ibrutinib
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
difference in microbiome biomarkers between patients developing colitis after exposure to targeted therapy and those not developing colitis | At the end of the study, after 2 years.
  With the different species and metabolites between the 2 groups of patients (patients developing diarrhea after exposure to Ibrutinib and those not developing diarrhea), we will create a risk score for occurrence of diarrhea during treatment with Ibrutinib, on the previously developed model (Montassier et al, 2016, Genome medicine)

SECONDARY OUTCOMES:
Identify biomarkers of the gut microbiota associated with the occurrence of severe diarrhea (grade 3 and 4 CTCAE, version 4.0) in patients treated with Ibrutinib for malignant hemopathy B. | At the end of the study, after 2 years.
Identify biomarkers of gut microbiota associated with the occurrence of diarrhea by subgroup: patients treated with Ibrutinib alone, patients treated with Ibrutinib in combination with another molecule | At the end of the study, after 2 years.
Creation of a predictive score of the occurrence of diarrhea in patients treated with Ibrutinib for malignant hemopathy B, including the biomarkers of the intestinal microbiome and the clinical characteristics of the patient | At the end of the study, after 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France